CLINICAL TRIAL: NCT00261287
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Clinical Trial Designed to Assess the Safety and Tolerability of Ciclesonide (200 mcg Once Daily), Applied as a Nasal Spray for Twelve Weeks, in the Treatment of Perennial Allergic Rhinitis (PAR) in Pediatric Patients 2-5 Years of Age
Brief Title: Safety and Tolerability of Ciclesonide Nasal Spray in Patients With Perennial Allergic Rhinitis (2-5 Years Old) (BY9010/M1-416)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-416
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: Hay Fever; Perennial Allergic Rhinitis
Keywords: Hay Fever; Allergic Rhinitis; Perennial Allergic Rhinitis; Ciclesonide
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic, Perennial; Rhinitis, Allergic | interventions — ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of ciclesonide nasal spray for long term use in relieving symptoms in perennial allergic rhinitis.

ELIGIBILITY:
Main Inclusion Criteria:

* General good health, other than perennial allergic rhinitis
* History and diagnosis of perennial allergic rhinitis by skin prick test
* History of perennial allergic rhinitis for a minimum of 90 days immediately before the screening visit

Main Exclusion Criteria:

* Participation in any investigational drug trial within the 30 days before the screening visit
* Use of any disallowed concomitant medications within the prescribed withdrawal periods before the screening visit
* A known hypersensitivity to any corticosteroid

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102
Dates: Start 2005-11; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ciclesonide nasal spray

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (3):
- United States (3):
  - Altana Pharma/Nycomed, Long Beach, California
  - Altana Pharma/Nycomed, Normal, Illinois
  - Altana Pharma/Nycomed, San Antonio, Texas

REFERENCES:
- See also: BY9010-M1-416-RDS-2007-03-22.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4539&filename=BY9010-M1-416-RDS-2007-03-22.pdf